CLINICAL TRIAL: NCT00002946
Title: A Phase I Trial of Oral Penclomedine
Brief Title: Penclomedine in Treating Patients With Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065413; WCCC-CO-9693; NCI-T96-0067; CDR0000065413 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-09-03 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-01

CONDITIONS: Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; unspecified adult solid tumor, protocol specific; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — penclomedine

ARMS (1):
- Arm I (Experimental): atients enrolled on the bioavailability portion of this study receive one dose of IV penclomedine over 1 hour followed by 2 weeks of rest. At the end of two weeks, they receive oral penclomedine for 5 days every 28 days. The starting dose is determined by a single primary patient who has been administered oral penclomedine and observed for dose limiting toxicity (DLT). [Bioavailability portion completed as of 3/98.] Those not on the bioavailability portion of study start on a standard design dose escalating schedule in which patients enroll in cohorts of 3. Patients are administered oral penclomedine daily for 5 days. This treatment repeats every 4 weeks. The MTD is defined as the dose immediately below that at which 2 patients experience DLT. Treatment repeats for 6 courses or until severe toxicity or tumor progression is observed.
  Interventions: Drug: penclomedine

INTERVENTIONS:
Drug: penclomedine

SUMMARY:
Phase I trial to study the effectiveness of penclomedine in treating patients with malignant solid tumors or lymphomas. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) and Phase II dose of oral penclomedine in patients with malignancies.

II. Determine the toxic effects of oral penclomedine in these patients. III. Determine the pharmacokinetics of oral penclomedine in these patients. IV. Determine the bioavailability of oral penclomedine in these patients.

OUTLINE:

Patients enrolled on the bioavailability portion of this study receive one dose of IV penclomedine over 1 hour followed by 2 weeks of rest. At the end of two weeks, they receive oral penclomedine for 5 days every 28 days. The starting dose is determined by a single primary patient who has been administered oral penclomedine and observed for dose limiting toxicity (DLT). [Bioavailability portion completed as of 3/98.] Those not on the bioavailability portion of study start on a standard design dose escalating schedule in which patients enroll in cohorts of 3. Patients are administered oral penclomedine daily for 5 days. This treatment repeats every 4 weeks. The MTD is defined as the dose immediately below that at which 2 patients experience DLT. Treatment repeats for 6 courses or until severe toxicity or tumor progression is observed.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy (solid tumor or lymphoma)
* No history of brain metastases

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Life expectancy: At least 12 weeks
* Performance status: ECOG 0-2
* WBC at least 4,000/mm3
* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Bilirubin less than 1.5 mg/dL
* Creatinine normal
* No history of seizure disorder Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior chemotherapy (6 weeks since nitrosoureas and mitomycin) and recovered
* At least 4 weeks since prior radiotherapy and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1997-10; Primary Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Wilding, MD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin, United States